CLINICAL TRIAL: NCT03176160
Title: Laser Interstitial Thermal Therapy (LITT) as Palliative Treatment for Patients With Malignant Glioma Requiring Standard Treatment Alternatives
Brief Title: LITT Palliative Treatment for Patients With Malignant Gliomas
Status: Withdrawn | Type: Observational
Why Stopped: Failure to enroll
Sponsor: Duke University (Other)
Collaborators: Monteris Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00079623
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Malignant Glioma of Brain; Glioblastoma
Keywords: LITT; Fecci; Pro00079623; Glioblastoma; Laser Interstitial Thermal Therapy; Palliative
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving palliative regimen consisting of LITT: Patients with WHO grade IV malignant glioma who are approved for and receive the LITT (Laser Interstitial Thermal Therapy) procedure
  Interventions: Other: Palliative regimen consisting of LITT

INTERVENTIONS:
Other: Palliative regimen consisting of LITT — Minimally invasive technique to necrotize intracranial lesions
  Other Names: NBS NeuroBlate® System

SUMMARY:
The purpose of this study is to to describe the effect of a palliative regimen consisting of Laser Interstitial Thermal Therapy (LITT) on distress, quality of life (QOL), neurocognition, days in the hospital, patient disposition, and readmission in newly diagnosed World Health Organization (WHO) grade IV malignant glioma (glioblastoma (GBM) or gliosarcoma) patients unable to undergo broader surgical resection. The primary objective is to assess changes in the National Comprehensive Cancer Network (NCCN) distress thermometer in newly diagnosed WHO grade IV malignant glioma patients who receive LITT.

*Please note: This study was originally designed as a interventional device study studying the effect of the LITT procedure; however, it was re-designed as an observational study in which the patient population being studied is approved to receive the LITT procedure.

DETAILED DESCRIPTION:
Patients will be identified from those previously approved for the LITT procedure. Following consent, 20 patients will complete NCCN distress, Quality of Life (QOL) and neuro-cognitive baseline testing, followed by the LITT procedure using the NeuroBlate® System (NBS) and intra-operative magnetic resonance imaging (MRI). Per standard clinical practice, after completing LITT, patients will undergo radiation at the discretion of the treating radiation oncologist. Patients will likewise receive concomitant and adjuvant chemotherapy (typically temozolomide) at the discretion of the treating neuro-oncologist. All patients will complete NCCN distress, QOL and neurocognitive testing immediately after the LITT procedure on post-operative day 1 as able, or immediately prior to discharge if more appropriate. Additionally, they will complete these same tests approximately 1, 3, 6, 12, and 24 months after the completion of LITT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histopathologically confirmed newly diagnosed WHO grade IV malignant glioma (GBM or gliosarcoma, multifocal disease is allowed) unable to undergo surgical resection, who is approved and scheduled to receive the LITT procedure by the treating neurosurgeon
* ≥18 years of age
* Patient is "fragile" (age 18-69, KPS 50-70), "elderly" (age > 69, KPS 80-100), or "elderly and fragile" (age > 69, KPS 50-70)
* Patient must not have received prior chemotherapy or brain radiotherapy
* Patient is able and willing to complete the QOL and neurocognitive questionnaires. Inability (illiteracy, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. If patients are not able to read or write, proxy interviews will be conducted in-person or via telephone by the assigned study clinician or study team member (Trail-Making A & B will not be performed on these patients).
* Patient consent must be obtained according to Duke institutional policy
* Patient must be accessible for follow-up

Exclusion Criteria:

* Non-English speaking or inability to read and understand English
* Patients with concurrent malignancies requiring active treatment, except: non-melanoma skin cancer, or in-situ cancer of the cervix.
* Patients with a serious active infection or other serious underlying medical conditions that would impair the ability of the patient to complete the protocol-related QOL and distress questionnaires and cognition assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed WHO grade IV malignant glioma who are unable to undergo broader surgical resection and are identified as approved to receive the LITT procedure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in NCCN distress thermometer score | Up to 24 months after the LITT procedure
  Mean change from baseline in the NCCN distress thermometer score

SECONDARY OUTCOMES:
Median overall survival | 24 months after LITT
  Overall survival will be defined as the time in months between Laser Interstitial Thermal Therapy (LITT) and death, or last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Change in Karnofsky Performance Status (KPS) | Up to 24 months after the LITT procedure
  Mean change from baseline in KPS score

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Fecci, MD, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/clinical-trials